CLINICAL TRIAL: NCT06026657
Title: Phase 1b/2 Study of Naxitamab (Danyelza), Gemcitabine and Ex Vivo Expanded Allogenic Universal Donor, TGFβi Natural Killer (NK) Cells in Advanced GD2-expressing Breast Cancers (DiG NKs)
Brief Title: Gemcitabine and Ex Vivo Expanded Allogenic Universal Donor, TGFβi Natural Killer (NK) Cells With or Without Naxitamab (Danyelza) for the Treatment of Patients With Metastatic, GD2 Expressing, HER2 Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Margaret Gatti-Mays (Other)
Responsible Party: Sponsor-Investigator, Margaret Gatti-Mays, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OSU-22237; NCI-2023-06508 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; HER2-Negative Breast Carcinoma
MeSH Terms: interventions — Specimen Handling; Gemcitabine; Magnetic Resonance Spectroscopy; naxitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm I (Gemcitabine, TGFBi) (Experimental): Patients receive gemcitabine intravenously (IV) over 30 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive TGFBi NK cells IV over 10-30 minutes on day 16 of cycle 1. Patients undergo CT scan and blood sample collection and may undergo MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Biological: Universal Donor Expanded TGF-beta-imprinted NK Cells
- Arm II (Gemcitabine, TGFBi x2) (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive TGFBi NK cells IV over 10-30 minutes on day 16 and 18 of cycle 1. Patients undergo CT scan and blood sample collection and may undergo MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Biological: Universal Donor Expanded TGF-beta-imprinted NK Cells
- Arm III (Gemcitabine naxitamab, TGFBi) (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 of each cycle followed by naxitamab IV over 30-60 minutes on days 1, 4, and 8 of each cycle. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive TGFBi NK cells IV over 10-30 minutes on day 16 of cycle 1. Patients undergo CT scan and blood sample collection and may undergo MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Biological: Naxitamab; Biological: Universal Donor Expanded TGF-beta-imprinted NK Cells
- Arm IV (Gemcitabine, naxitamab, TGFBi x2) (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 of each cycle followed by naxitamab IV over 30-60 minutes on days 1, 4, and 8 of each cycle. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive TGFBi NK cells IV over 10-30 minutes on day 16 and 18 of cycle 1. Patients undergo CT scan and blood sample collection and may undergo MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Biological: Naxitamab; Biological: Universal Donor Expanded TGF-beta-imprinted NK Cells

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Naxitamab — Given IV
  Other Names: Anti-Gd2 IGG3 Monoclonal Antibody 3f8 Humanized; Danyelza; Hu3F8; Humanized Anti-GD2 Antibody 3F8; Humanized Monoclonal Antibody Hu3f8-IGG1
  Arms: Arm III (Gemcitabine naxitamab, TGFBi); Arm IV (Gemcitabine, naxitamab, TGFBi x2)
Biological: Universal Donor Expanded TGF-beta-imprinted NK Cells — Given IV
  Other Names: Allogeneic TGFBi Expanded NK Cells; UD TGF-betai NK Cells; Universal Donor TGF-beta Imprinted Expanded NK Cells

SUMMARY:
This phase Ib/II trial tests the safety, best dose and how well gemcitabine and ex vivo expanded allogenic universal donor TGFBi NK cells with or without naxitamab work for the treatment of patients with GD2 expressing, HER2 negative breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Gemcitabine is a chemotherapy drug that blocks the cells from making deoxyribonucleic acid (DNA) and may kill cancer cells. TGFBi NK cells are manufactured cells that are a part of your natural immunity. NK cells can recognize missing or incorrect proteins on tumor cells and then eliminate these tumor cells and TGFBi NK cells are created to be able to better kill the tumor cells. Naxitamab is a monoclonal antibody that targets GD2, which is a protein or sugar present on tumor cells but not very commonly found on normal cells. This antibody helps draw the attention of the immune system to the tumor cells that have GD2 to help attack the tumor cells. Giving gemcitabine and TGFBi NK cells with or without naxitamab may kill more tumor cells in patients with metastatic GD2 expressing, HER2 negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of gemcitabine plus transforming growth factor beta imprinted natural killer (TGFBi NKs) +/- naxitamab in metastatic breast cancer.

II. To evaluate the objective response rate of gemcitabine plus TGFB NKs +/- naxitamab in metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To determine if TGFB NK cells are detectable in the peripheral blood 5 days following infusion (C1D21).

II. To determine if gemcitabine plus TGFB NKs +/- naxitamab improves median progression-free survival (PFS) in metastatic breast cancer over historical controls for gemcitabine alone.

EXPLORATORY OBJECTIVES:

I. Peripheral blood mononuclear cells (PBMCs) Ia. Real-time blood immune profiling Ib. Antigen specific immune responses II. Plasma/Serum IIa. TCR clonality IIb. Cytokines (IFNy, IL-10, IL-12, IL-2, IL4, etc) and chemokines IIc. Antigen specific immune responses III. Archival tissue IIIa. GD2 expression on tumor IIIb. Immunohistochemistry/multispectral imaging IIIc. Tumor mutational burden

OUTLINE: Patients are assigned to 1 of 4 arms.

ARM I: Patients receive gemcitabine intravenously (IV) over 30 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive TGFBi NK cells IV over 10-30 minutes on day 16 of cycle 1.

ARM II: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive TGFBi NK cells IV over 10-30 minutes on day 16 and 18 of cycle 1.

ARM III: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 of each cycle followed by naxitamab IV over 30-60 minutes on days 1, 4, and 8 of each cycle. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive TGFBi NK cells IV over 10-30 minutes on day 16 of cycle 1.

ARM IV: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 of each cycle followed by naxitamab IV over 30-60 minutes on days 1, 4, and 8 of each cycle. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive TGFBi NK cells IV over 10-30 minutes on day 16 and 18 of cycle 1.

Patients undergo computed tomography and blood sample collection and may undergo magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up within 30 days of stopping treatment and every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed, HER2 negative metastatic breast cancer that is historically GD2 expressing (e.g., triple negative breast cancer, metaplastic breast cancer, high grade 3 estrogen positive breast cancer at initial diagnosis) with available archival tissue. Well differentiated neuroendocrine tumor (NETs) are not eligible for this trial since GD2 expression is unknown. GD2 expression is not required for eligibility but a primary tumor paraffin block is required at enrollment for assessment of GD2 expression
* Patients must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for the evaluation of measurable disease
* Patients must have received at least one prior treatment for metastatic disease and progressed on treatment or been intolerant to treatment
* Female or male >=18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count >= 1,500/mcL (> 1.5 X 10^6/L)
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 mg/dL (transfusion to obtain hemoglobin >= 9 mg/dL within 24 hours prior to dosing is allowed)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) or measured or calculated creatinine clearance (CrCl) >= 60 mL/min for participant with creatinine levels > 1.5 X institutional upper limit of normal (ULN) (Glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl)
* Patients must have adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels =< 3 X ULN and total bilirubin < 1.5 X ULN, unless known diagnosis of Gilbert's syndrome, where bilirubin =< 5 mg/dL will be permitted. Gilbert's syndrome will be defined as elevated unconjugated bilirubin, with conjugated (direct) bilirubin within the normal range and less than 20% of the total. Total bilirubin will be permitted up to 5 mg/dL, if patients have historical readings consistent with the definition of Gilbert's syndrome prior to entering study. Adequate hepatic function for patients with known liver metastases is defined as AST and ALT levels ≤ 5 X ULN
* The effects of the trial agents on the developing human fetus are unknown. However, gemcitabine is known to have negative fetal effects. For this reason: Women of childbearing potential must agree to use adequate contraception at study entry, for the duration of study participation and for 7 months after the last dose of study medication based upon estimated half-life or receptor occupancy. Adequate contraception is defined as 2 highly effective methods of contraception (including a physical barrier). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men should refrain from fathering a child using adequate contraception or donating sperm during the study and for 6 months after the last dose of study medications. Adequate contraception is defined as 2 highly effective methods of contraception (including a physical barrier)
* Patients with well-controlled human immunodeficiency virus (HIV) infection are eligible for trial as long as:

  * On an effective anti-retroviral therapy (ART) ˃ 4 weeks and with evidence of viral-suppression as defined as HIV viral load ˂ 400 copies/mL within the last 3 months
  * CD4 > 200 cells/µL within the last 3 months; and
  * No reported opportunistic infections within 6 months prior to enrollment, except for the following which will be allowed:

    * Esophageal candidiasis treated within last 6 months or currently improving with antifungal treatment.
    * Oral and/or genital herpes simplex virus (HSV) treated within last 6 months or currently improving with antiviral treatment.
    * Mycobacterium avium infection in last 6 months or that has been treated for at least 1 month
* Patients with evidence of chronic hepatitis B virus (HBV) infection are eligible for trial as long as the HBV viral load is undetectable on suppressive therapy, if indicated.

  * Patients with history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable or unquantifiable HCV ribonucleic acid (RNA) 12 weeks or longer after definitive treatment completion.
  * Patients must be able to understand and willing to sign a written informed consent document
* Any adverse events subjects have experienced from prior therapy must have resolved to =< grade 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5

Exclusion Criteria:

* Patients who within 3 weeks prior to study enrollment who have received chemotherapy, investigational agents, or radiation
* Patients with active brain metastases or leptomeningeal metastases are excluded from this clinical trial because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients with treated brain metastases are eligible if there is no magnetic resonance imaging (MRI) evidence of progression for 6 months after treatment is complete and within 28 days prior to the first dose of trial drug. Patients requiring immunosuppressive doses of systemic corticosteroids (> 10mg/day prednisone equivalent) for palliation are excluded
* Patients with a history of another invasive malignancy < 3 years prior to enrollment (patients with non-melanoma skin cancers, carcinoma in situ of the breast or cervix are eligible)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection that requires systemic treatment with ongoing antibiotics (eligible if can stop antibiotics on day of enrollment), unexplained fever (temperature > 38.1˚celcius [C]) within 7 days of initial treatment, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that in the opinion of the primary investigator would prohibit the patient from complying with study requirements
* Patients with bone metastases who have initiated denosumab or a bisphosphonate therapy within 28 days prior to or after cycle 1 day 1 due to the potential for flu-like symptoms and mild cytokine release syndrome with the initial dose. However, continuation of prior therapy is allowed
* Patients should have no evidence of being immunocompromised as listed below:

  * Active, known or suspected autoimmune disease. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to an autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger in the opinion of the primary investigator
  * Altered immune function that in the judgement of the PI that may affect a patient's ability to adequately engage the immune system and respond to the immunotherapy agents being administered, including but not limited to: inflammatory bowel disease; active infectious enteritis; eosinophilic enteritis; lupus erythematous; ankylosing spondylitis; scleroderma; multiple sclerosis. These criteria do not include all disease with an immune-related component but are not autoimmune in nature or have a primary alteration in the general immune function that may interfere with the vaccine mechanism of action, for example celiac disease
  * Immunosuppressive therapy post-organ transplant
  * Concurrent use of chronic use of systemic steroids, except for physiologic doses of systemic steroids for replacement, defined as 10mg of prednisone per day or equivalent, or local (topical, nasal, ophthalmic or inhaled) steroid use or prior concomitant use with chemotherapy. Systemic steroids must have been discontinued >2 weeks prior to trial start. Prior use of corticosteroids in short-term schemes (duration shorter than 3 days) for indications such as prophylaxis of reactions to intravenous contrast for imaging studies or chemotherapy-related adverse events (AEs) are not considered part of this exclusion. Prior use of corticosteroids for brain metastasis ending at least 14 days prior to enrollment is not considered part of this exclusion criteria
* Pregnant and breastfeeding women are excluded from this study because of the potential for teratogenic or abortifacient effects with all of the agents involved in this trial. Females of childbearing potential who are pregnant, breast feeding, intend to become pregnant, or are not using adequate contraceptive methods or males who are not using adequate contraceptive methods. Women of childbearing potential must agree to use two methods of adequate contraception at study entry be used for the duration of study participation and for at least 7 months for women and 6 months for men after the final dose of any study-related medications
* Clinically significant cardiomyopathy, coronary disease, myocardial infarction, chronic heart failure (CHF) (New York Heart Association class III or IV or hospitalization for CHF), ejection fraction < 50% or cerebrovascular accident within 6 months prior to enrollment
* Patients with a history of myocarditis are excluded due to the potential of myocarditis with anti-PD-L1 antibodies or other immunotherapies
* Patients who have received any live vaccines within 30 days prior to enrollment (inactivated vaccines including COVID vaccines are allowed)
* Any other condition, which would, in the opinion of the principal investigator the subject is a poor candidate for the clinical trial or would jeopardize the subject or the integrity of the data obtained
* Inadequate pulmonary function defined as evidence of dyspnea at rest, exercise intolerance, and/or chronic oxygen requirement. In addition, room air pulse oximetry < 90% and/or abnormal pulmonary function tests within 28 days of C1D1 if these assessments are clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 year after completion of study medication
  Will be summarized descriptively with reporting of any dose limiting toxicities (DLTs) in these initial patients. In addition, to DLTs, serious adverse events (SAEs) and immune related adverse events of interest will be reported. Will be summarized descriptively and graphically, with reporting the outcome measures indicated along with two-tailed 95% confidence intervals (CIs). Number and frequency of patients experiencing each adverse event (AE) type and grade will tabulated, among patients evaluable for toxicity. The number (%) of patients experiencing at least one grade 3 to 5 AE will be reported with 95% CI.
Objective response rate | Up to 1 year after completion of study medication
  Will be estimated in each arm using two-sided 80% and 95% CI about the observed percentages of response (PR+CR).

SECONDARY OUTCOMES:
Transforming growth factor beta imprinted natural killer (TGFBi NK) cell detection | At day 5 following infusion
  TGFBi NK cell persistence will be defined as the presence (detectable donor TGFBi NK cells) or the absence (no detectable donor TGFBi NK cells). Data will be described numerically as percentage of donor cells in blood and will be correlated to clinical outcomes.
Progression free survival | From start of treatment to time of progression or death, whichever occurs first, up to 1 year after completion of study medication
  Will be estimated using a Kaplan-Meier curve and the median PFS will be reported along with a 95% confidence interval, separately by arm, based on the patients who are enrolled in the evaluation of clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E Gatti-Mays, MD MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu